CLINICAL TRIAL: NCT00876577
Title: VICTOR - Avelox® i.v. in Acute Exacerbations of Chronic Bronchitis
Brief Title: VICTOR - Avelox® Intravenous (i.v.) in Acute Exacerbations of Chronic Bronchitis
Acronym: VICTOR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Healthcare AG
Other Study IDs: 14495; AX0810CN (Other: Company internal)
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Bronchitis; Disease Exacerbation
Keywords: Acute Exacerbations of Chronic Bronchitis; Avelox; Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic; Disease Progression; Bronchitis | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Patients from the normal praxis routine, treated with Moxifloxacin injection with/without sequential tablet treatment according to the local product information

SUMMARY:
This study is a local, prospective, open-label, company-sponsored, non interventional, multi-center study. Patients documented must suffer from an acute exacerbation of chronic bronchitis and take at least one dose of Moxifloxacin injection.The primary objective is to obtain clinical effectiveness and safety data of Moxifloxacin injection in the treatment of acute exacerbations of chronic bronchitis in patients in whom Moxifloxacin was routinely prescribed. The secondary objective is to find out the possible correlation between the risk factors (sex, smoking, number of previous exacerbations, etc) and AECB, the different treatment effectiveness according to Anthonisen classification. This study will also collect the data of pathogens by sputum culture and the defervescence time of Moxifloxacin injection in treating Acute Exacerbations of Chronic Bronchitis (AECB).

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age with a diagnosis of AECB treated with Moxifloxacin injection with/without sequential tablet treatment

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with AECB, who are at least 18 years of age and are scheduled to be treated with Moxifloxacin injection, independent of the duration and severity of the underlying chronic bronchitis, can be documented after the therapy decision has been made.
Sampling Method: Non-Probability Sample
Enrollment: 1206 (Actual)
Dates: Start 2009-05; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
clinical cure rate:clinical cure was defined as disappearance of acute signs and symptoms | up to 21 days

SECONDARY OUTCOMES:
Time to cure: time when symptoms are disappeared after Moxifloxacin treatment | up to 21 days
Improvement time: time when patients feel improvemen | up to 21 days
Time of patients recover from fever | up to 21 days
Clinical efficacy rate of Moxifloxacin | up to 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, China